CLINICAL TRIAL: NCT02632825
Title: Effects of Nasal High Flow Therapy on Ventilation and Gas Exchange During Wakefulness and Sleep in Healthy Newborn Babies in a Randomized Crossover Study Design
Brief Title: Effects of Nasal High Flow Therapy on Ventilation and Gas Exchange in Healthy Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Center of Maternal and Child Health Protection, Armenia (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RCMCHP014
Record Dates: First submitted 2015-09-10; First posted 2015-12-17 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Support
Keywords: Nasal High Flow; gas exchange; newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal High Flow (Experimental): NHF will be applied at 8 L/min (AIRVO 2) through (OPT 316) Optiflow nasal cannula interface without supplemental oxygen
  Interventions: Device: Nasal High Flow
- Control (No Intervention): Control is no NHF intervention

INTERVENTIONS:
Device: Nasal High Flow — Nasal High Flow Therapy
  Arms: Nasal High Flow

SUMMARY:
Nasal High Flow (NHF) and CPAP are established forms of respiratory support in neonates and often produce similar clinical outcomes. It has been shown in adults that NHF produce different effects on ventilation during wakefulness and sleep. There is no physiological data on effects of NHF in neonates. The physiological effects may be impacted by sleep/awake status.

DETAILED DESCRIPTION:
The aim of the study to investigate the effects of NHF therapy on ventilation and gas exchange during wakefulness and sleep in healthy term newborns.

Interventions:

NHF will be applied at 8 L/min (AIRVO 2) via (OPT 316) Optiflow nasal cannula interface without supplemental oxygen. Participants will act as their own control (no intervention) in a randomized crossover study design.

Physiological measurements:

1. Ventilation will be assessed using Respiratory Inductance Plethysmography (RIP) (Respitrace QDC, Viasys, USA).
2. Blood carbon dioxide (CO2) and oxygen levels will be measured by a non-invasive transcutaneous monitor (Tosca, Radiometer, Demnark).
3. All experiment will be recorded using Analogue-to-Digital converter (Powerlab, ADInstruments, New Zealand) and LabChart software with video recording of the patient.
4. Sleep/awake statuss will be determined by videorecording of the patient and Electroencephalogram (EEG) (Alice Polysomnography System Philips, USA)
5. The total study time will be <3 hours in total for each participant. Routine measurement of heart rate, respiratory rate and oxygen saturation will be performed as per standard neonatal clinical practice.
6. Intervention can be terminated if at any time SpO2 drops below 80%, TcCO2 increases above 60 mm Hg, Respiratory Rate increases above 80 breaths per min for more than one minute).

The researcher is an experienced neonatal consultant will be conducting the research and observing the baby throughout the study.

Protocol:

Both control and NHF intervention periods will last a maximum of 40 min each. The maximum duration of the study including set-up, calibration, intervention, washout ans control will be <3 hours. At the beginning of the study when all probes are attached a self-calibration period of RIP will be followed by a calibration of breathing volume with a pneumotachometer attached to a nasal mask. After all calibrations are completed a baseline measurement will be followed by either NHF 8 L/min or a control period without NHF. At the end of this period the interventions will be changes either to control or NHF, which will follow by a washout period (no NHF) and an additional calibration of RIP with a pneumotachometer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy full or near full-term newborns of 1-2 days of age.
* A parent has given written informed consent to their baby's participation.

Exclusion Criteria:

* Infants who are clinically unstable and unsuitable for non-invasive respiratory support as judged by consultant clinician or required supplemental oxygen.
* Known upper airway, lower respiratory tract, cardiac or gastrointestinal tract anomaly.
* A parent has not given written informed consent.

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change of minute ventilation | Up to 1 hour
  Change of minute ventilation measured with calibrated Respiratory Inductance Plethysmography
Change of respiratory rate | Up to 1 hour
  Change of respiratory rate measured with Respiratory Inductance Plethysmography

SECONDARY OUTCOMES:
Tissue carbon dioxide | Up to 1 hour
  Change of transcutaneous tissue carbon dioxide
Tissue oxygen | Up to 1 hour
  Change of transcutaneous oxygen
Oxygen saturation | Up to 1 hour
  SpO2
Heart rate | Up to 1 hour
  Heart rate measured with pulseoximeter

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Mazmanyan, MD, PhD, Principal Investigator — Head of Neonatal Unit of Research Centre of Maternal and Child Health
Locations (1):
- Neonatal Intensive Care Unit, Research Centre of Maternal and Child Health, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No